CLINICAL TRIAL: NCT07296705
Title: Selective Bladder Preservation After Neoadjuvant Zanidatamab Combined With Tislelizumab and Chemotherapy in Patients With HER2-Positive Muscle-Invasive Bladder Cancer: A Multicenter Study
Brief Title: Neoadjuvant Zanidatamab + Tislelizumab + Chemotherapy for Selective Bladder Preservation in HER2-Positive MIBC
Acronym: HARBOR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Medical University Union Hospital (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HARBOR-II-2025
Record Dates: First submitted 2025-09-26; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-09

CONDITIONS: Muscle Invasive Bladder Cancer (MIBC)
MeSH Terms: interventions — zanidatamab; tislelizumab; Cisplatin; Gemcitabine; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: Zanidatamab; Drug: Tislelizumab; Drug: Cisplatin; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Zanidatamab — Zanidatamab (1,800 mg for patients <70 kg or 2,400 mg for patients ≥70 kg, administered intravenously every 3 weeks) for 4 cycles is given as part of the neoadjuvant regimen. After completion of neoadjuvant therapy, disease status is reassessed. Patients achieving a clinical complete response (cCR) may continue zanidatamab every 3 weeks for 2-4 cycles as part of bladder-preserving treatment; those without cCR may receive radiotherapy or partial cystectomy followed by zanidatamab every 3 weeks for 2-4 cycles, or undergo radical cystectomy without further zanidatamab treatment.
Drug: Tislelizumab — Tislelizumab (200 mg administered intravenously every 3 weeks) is administered for 4 cycles as neoadjuvant therapy. After completion of 4 cycles, disease status is reassessed. Patients achieving a clinical complete response (cCR) may proceed with selective bladder preservation and continue tislelizumab every 3 weeks for 12 cycles; those without cCR may receive radiotherapy or partial cystectomy followed by tislelizumab every 3 weeks for 12 cycles, or undergo radical cystectomy with adjuvant tislelizumab every 3 weeks for 12 cycles.
Drug: Cisplatin — Cisplatin (70 mg/m² administered intravenously every 3 weeks ) for 4 cycles is included in the neoadjuvant chemotherapy regimen for eligible cisplatin-based chemotherapy.
Drug: Gemcitabine — Gemcitabine (1,000 mg/m² administered intravenously every 3 weeks) for 4 cycles is given as part of the neoadjuvant chemotherapy regimen for eligible cisplatin-based chemotherapy.
Drug: Nab-paclitaxel — Nab-paclitaxel (125 mg/m² administered intravenously every 3 weeks) for 4 cycles is given as part of the neoadjuvant chemotherapy regimen for ineligible or refused cisplatin-based chemotherapy.

SUMMARY:
This is a multicenter, open-label, prospective, single-arm, phase II study designed to evaluate the efficacy and safety of neoadjuvant zanidatamab combined with tislelizumab and chemotherapy, followed by selective bladder preservation, in patients with HER2-positive muscle-invasive bladder cancer (MIBC) staged cT2-4aN0-1M0.

DETAILED DESCRIPTION:
Eligible patients will receive neoadjuvant therapy with zanidatamab plus tislelizumab in combination with chemotherapy, followed by clinical reassessment. Patients who achieve a clinical complete response (cCR) will continue maintenance therapy with zanidatamab and tislelizumab. Patients who do not achieve cCR may, undergo radiotherapy or partial cystectomy and then continue maintenance zanidatamab plus tislelizumab; alternatively, they may proceed directly to radical cystectomy followed by adjuvant tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate, able to provide written informed consent, and able to understand and comply with study requirements and the assessment schedule.
2. Age 18 to 85 years on the date of informed consent.
3. Residual disease after TURBT; histologically confirmed urothelial carcinoma of the bladder staged cT2-T4aN0-1M0 per AJCC 8th edition by histology and imaging. For mixed histology, urothelial carcinoma must be predominant (≥50%).
4. Availability of TURBT tumor tissue and corresponding pathology report; either fresh surgical tissue or unstained slides may be submitted.
5. HER2-positive: IHC 2+ or 3+.
6. No prior anti-HER2-directed therapy (including but not limited to HER2 antibodies, HER2-targeting ADCs, or HER2-targeted TKIs) and no prior PD-(L)1 therapy.
7. ECOG performance status 0-2.
8. Adequate organ function based on screening labs obtained ≤14 days before enrollment:

   a. For the following counts, no growth-factor support within 14 days prior to sample collection: i. Absolute neutrophil count ≥ 1.5 × 10^9/L ii. Platelets ≥ 100 × 10^9/L iii. Hemoglobin ≥ 90 g/L b. INR or aPTT ≤ 1.5 × upper limit of normal (ULN) c. Total bilirubin ≤ 1.5 × ULN (≤ 3 × ULN for Gilbert syndrome or isolated indirect hyperbilirubinemia) d. AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN
9. Women of childbearing potential must have a negative urine or serum pregnancy test within ≤7 days before enrollment and agree to use highly effective contraception during the study and for ≥120 days after the last dose of zanidatamab, tislelizumab, or chemotherapy (whichever occurs later).
10. Non-sterilized men must agree to use highly effective contraception during the study and for ≥120 days after the last dose of zanidatamab, tislelizumab, or chemotherapy (whichever occurs later).

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Uncontrolled infection requiring systemic therapy.
3. Diagnosis of another malignancy within the past 5 years.
4. Major surgery or significant trauma within 28 days prior to enrollment (placement of a vascular access device and TURBT are not considered major surgery).
5. Prior radiotherapy to the bladder for bladder cancer.
6. Active autoimmune disease requiring systemic treatment that, in the investigator's judgment, would affect study therapy.
7. Any of the following cardiovascular criteria:

   1. Cardiac chest pain within ≤28 days before first study dose, defined as moderate pain that limits activities of daily living.
   2. Symptomatic pulmonary embolism within ≤28 days before first study dose.
   3. Any acute myocardial infarction within ≤6 months before first study dose.
   4. Any history of heart failure of New York Heart Association (NYHA) Class III or IV within ≤6 months before first study dose.
   5. Any ventricular arrhythmia of severity ≥ Grade 2 within ≤6 months before first study dose.
   6. Any cerebrovascular accident within ≤6 months before first study dose.
   7. Corrected QT interval (QTc by Fridericia): ≥470 msec for women or ≥450 msec for men.

   i. Note: If the initial ECG shows QTc >450 msec (men) or >470 msec (women), a follow-up ECG should be performed to confirm.

   h) Left ventricular ejection fraction (LVEF) ≤50% by multigated acquisition (MUGA) scan or echocardiography (ECHO). The same modality used at baseline must be used for follow-up assessments.
8. History of acute myocardial infarction or ischemic stroke within 6 months.
9. Human immunodeficiency virus (HIV) infection (i.e., positive antibodies to HIV-1/2), active syphilis infection, or active tuberculosis infection.
10. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
11. History of interstitial lung disease, non-infectious pneumonitis, or uncontrolled pulmonary disease, including pulmonary fibrosis or acute lung disease.
12. Known hypersensitivity to any study drug.
13. Concurrent participation in another clinical study, unless observational (non-interventional) or in the follow-up phase of an interventional study.
14. Any other condition deemed by the investigator to render the patient ineligible.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Complete Response (cCR) Rate | At the end of Cycle 4 of neoadjuvant therapy (each cycle is 21 days)
  Proportion of participants achieving cCR at the end of neoadjuvant therapy, defined as no evidence of tumor on radiographic imaging, no residual tumor on diagnostic TURBT, and negative urine cytology

SECONDARY OUTCOMES:
1-Year Bladder-Intact Disease-Free Survival (BI-DFS) | From first neoadjuvant dose to 12 months
  Percentage of participants who, within 12 months from the first neoadjuvant dose, have no local or regional recurrence, no distant metastasis, no bladder cancer-related death, and have not undergone radical cystectomy
2-Year Bladder-Intact Disease-Free Survival (BI-DFS) | From first neoadjuvant dose to 24 months
  Percentage of participants who, within 24 months from the first neoadjuvant dose, have no local or regional recurrence, no distant metastasis, no bladder cancer-related death, and have not undergone radical cystectomy
Local Recurrence Free Survival (LRFS) | From first neoadjuvant dose until event, assess up to 3 years
  Time from the first neoadjuvant dose to local recurrence or death from any cause; participants without an event will be censored at last follow-up
Distant Metastasis Free Survival (DMFS) | From first neoadjuvant dose until event, assess up to 3 years
  Time from the first neoadjuvant dose to distant metastasis or death from any cause; participants without an event will be censored at last follow-up
Overall Survival (OS) | From first neoadjuvant dose until death, assess up to 3 years
  Time from the first neoadjuvant dose to death from any cause; participants alive at analysis will be censored at last follow-up.
Safety and Adverse Events | From first dose through last follow-up, assess up to 3 years
  Summary of study drug exposure (duration and dose) and adverse events
Quality of Life Assessed by EORTC QLQ-C30 | From baseline through last follow-up, assess up to 3 years
  To assess changes in overall and cancer-specific quality of life (QoL) from baseline to post-treatment using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) in patients with HER2-positive MIBC receiving neoadjuvant and selective bladder-preserving therapy.
Quality of Life Assessed by FACT-BI | From baseline through last follow-up, assess up to 3 years
  To assess changes in bladder cancer-specific quality of life (QoL) from baseline to post-treatment using the Functional Assessment of Cancer Therapy-Bladder (FACT-BI) questionnaire in patients with HER2-positive MIBC receiving neoadjuvant and selective bladder-preserving therapy.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital Affiliated to Fuzhou University, Fuzhou, Fujian
  - Affiliated Hospital of Putian University, Putian, Fujian
  - Quanzhou First Hospital Affiliated to Fujian Medical University, Quanzhou, Fujian
  - Sanming First Hospital, Sanming, Fujian
  - The First Affi liated Hospital of Xiamen University, Xiamen, Fujian
  - Zhangzhou Affiliated Hospital to Fujian Medical University, Zhangzhou, Fujian
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No